CLINICAL TRIAL: NCT01026311
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Efficacy of Coenzyme Q10 in Improving Mitochondrial Function in Older Athletes Treated With Statin Medications
Brief Title: Coenzyme Q10 in Older Athletes Treated With Statin Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Richard Deichmann, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Deichmann, MD, PI, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 09-076
Record Dates: First submitted 2009-12-01; First posted 2009-12-04 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Muscle Weakness; Myalgia; Side Effects of Statins
Keywords: Coenzyme q10; statins; myalgias; anaerobic threshold; athletic performance
MeSH Terms: conditions — Muscle Weakness; Myalgia | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Coenzyme Q10 (Active Comparator): 200mg of coenzyme Q10
  Interventions: Drug: Coenzyme q 10

INTERVENTIONS:
Drug: Coenzyme q 10 — 200 mg of Coenzyme q 10
  Arms: Coenzyme Q10
Drug: placebo — 1 placebo q d during treatment period
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effect of coenzyme Q10 administration in improving mitochondrial function as measured by anaerobic threshold in older athletes on a stable dose of statin medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 50 years of age, male or female.
* Patients on a stable dose of statin medication for at least 3 months prior to enrollment in the study
* Self-Described Athletes with any of the following characteristics:

  * Participation in a competitive athletic event within the past year or currently training for a competitive athletic event within the 6 months following enrollment
  * Regular exercise activity of at least 45 minutes duration 5 times per week

Exclusion Criteria:

* Use of coenzyme Q10 during the preceding two months.
* CPK level at baseline greater than two times the upper limits of normal
* LDL level at baseline greater than 160 for those without a cardiovascular risk or cardiovascular risk equivalent
* LDL level at baseline greater than 130 for those with a cardiovascular risk or cardiovascular risk equivalent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to test if oral coenzyme Q10 is superior to placebo in improving oxygen consumption by mitochondria as measured by cardiopulmonary fitness testing for anaerobic threshold in this population | The study will consist of an initial six week treatment period followed by a six week washout period. Subjects will then crossover to the alternative treatment for a second six week study period.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Deichmann, MD, Principal Investigator — Ochsner
Locations (1):
- Ochsner, New Orleans, Louisiana, United States